CLINICAL TRIAL: NCT04256070
Title: Effect of Education and Tele-consultancy Intervention Based on Watson Human Care Theory on Self-efficacy and Quality of Life Individuals With COPD
Brief Title: Effect of Education and Tele-consultancy Intervention Based on Watson Human Care Theory Individuals With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Şehnaz Kaya, Principal investigator, PhD student, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2012-KAEK-20, Karar no: 718
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Self Efficacy; Quality of Life; Pulmonary Function; Nurse's Role
Keywords: chronic obstructive pulmonary disease; nursing; quality of life; self-efficacy; Watson's Human Care Theory
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education, tele-consultation and training booklet (Experimental): * Informed Consent Form will be taken in written from those who agree to participate in the research.
  * In the first intervention, Information Form Based on Watson's Human Care Theory, Chronic Obstructive Pulmonary Disease Self-efficacy Scale, St. George Quality of Life Scale, Respiratory Function Test Form data will be collected. Subsequently, education, counseling nursing care and education booklet based on Watson's Human Care Theory will be given.
  Teleconsultation based on Watson's Human Care Theory will be given during the intervention at weeks 2, 4, 6, 8 and 10.
  * 24-hour tele-consultancy will be given on subjects determined for the management of COPD in case of necessity at the request of the individual.
  * In the last intervention in the 12th week, face to face with the individual, Consultancy based on Watson Human Care Theory, Self-efficacy Scale, St. George Quality of Life Scale, Respiratory Function Test Form, Telephone Interview Evaluation Form will be applied.
  Interventions: Behavioral: education and tele-consultation
- Standart care, no intervention (No Intervention): * Informed Consent Form will be taken in writing from those who agree to participate in the research.
  * At the first meeting, Information Form Based on Watson Human Care Theory, Self-efficacy Scale, St. George Quality of Life Scale, Respiratory Function Test Form data will be collected.
  Interventions will not be applied to individuals in this group and routine treatment and follow-up will continue.
  - COPD Self-efficacy Scale, face-to-face meeting at the end of the 12th week. George Quality of Life Scale, Respiratory Function Test Form will be repeated.
  A training booklet for COPD management will be provided.

INTERVENTIONS:
Behavioral: education and tele-consultation — education and tele-consultation based on Watson's Human Care Theory
  Arms: Education, tele-consultation and training booklet

SUMMARY:
This study aims to investigate the effect of education and tele-consultancy intervention based on Watson's Human Care Theory on self-efficacy and quality of life of individuals with COPD.

DETAILED DESCRIPTION:
: The research that a single-blinded randomized controlled trial, a total of 74 individuals, including 37 individual intervention and 37 individual control groups who applied to Akdeniz University Chest Diseases Polyclinic for consultation and follow-up, meeting the inclusion criteria, conducted between October 2020 - May 2022. In collecting data Information Form Based on Watson Human Care Theory, the Chronic Obstructive Pulmonary Disease Self-efficacy Scale, St. George Quality of Life Scale, and Pulmonary Function Test Form were used. Individuals in the intervention group were provided with training and consultancy based on Watson Human Care Theory, and an educational booklet prepared with current guides and expert opinions. Telephone counseling was provided in the 2nd, 4th, 6th, 8th, and 10th weeks after the first intervention in the intervention group. Routine follow-up of individuals in the control group was continued. The data of the scales in the intervention and control groups are collected in the 12th week. The individuals in the control group were given a training booklet at the end of the study. Statistical analysis of the data was done with SPSS 22.0 software package.

ELIGIBILITY:
Inclusion Criteria:

* Who has been diagnosed with COPD for more than 6 months
* No exacerbation for at least 4 weeks, stable period
* Followed up at Akdeniz University Hospital Chest Diseases Polyclinic
* Clear conscious (evaluated by Sandartize Mini-Mental Test higher than 23 points)
* No verbal communication barriers
* Individual phone owner
* No hearing or communication problems on the phone
* 18 years and older
* Literate
* Agree to participate in the research

Exclusion Criteria:

* Not getting enough points from the Standardized Mini-Mental Test
* A diagnosis of malignancy (based on file information)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Chronic Obstructive Pulmonary Disease Self-Efficacy Scale | from baseline and at the end of the third months
  To measure self-efficacy in Chronic Obstructive Pulmonary Disease (COPD), Wigal et al. (1991) developed The Chronic Obstructive Pulmonary Disease Self-Efficacy Scale. The total score is calculated by the score of each of the answers given. There are 34 items in the total of the subtitles, a minimum of 34 points and a maximum of 170 points. High scores indicate that the level of self-efficacy is high. To find the overall score of the subscales, the total score is divided by the number of items that make up the subscale. In comparison, if there is an increase in score in the posttest compared to the pretest, it is interpreted that the degree of confidence in managing breathing difficulties or avoiding increased. By translating the scale into Turkish, Kara and Mirici (2002) tested its validity and reliability. Cronbach's alpha value in the original version of the scale is 0.95; Cronbach's alpha value of the Turkish version was found to be 0.94.

SECONDARY OUTCOMES:
St. George's Respiratory Questionnaire | from baseline and at the end of the third months
  St. George's Respiratory Questionnaire (SGRQ) is known to be associated with the most commonly used scales in respiratory diseases. SGRQ is a 50-item scale under three main titles developed in 2001: symptoms (8 items), activities (16 items), effects of the disease (26 items).
  It is a scale that investigates the relationship between dyspnea, sputum, cough, respiratory status, and daily activity, especially in individuals with COPD. Its highest score is 100 and it expresses the highest level of negative status. Cronbach's alpha value of SGRQ was calculated as 0.88 for the whole scale, and it was found in the validity analysis that it correlated significantly with similar scales (p <0.0001). The SGRQ scale was translated into Turkish by Polatlı et al. (2013) and its validity and reliability study was conducted. Correlation of Turkish version Cronbach's alpha value was found to be 0.90.

OTHER OUTCOMES:
Pulmonary function tests | from baseline and at the end of the third months
  It is known that spirometry is the best method in the evaluation of airway obstruction and COPD. After spirometry, forced vital capacity (FVC), forced expiration volume in 1 second (FEV1), FEV1 / FVC ratio values are obtained. Normal values of the FEV1 / FVC ratio between 0.7-0.8 and less than 0.65 are indicative of airway obstruction. After spirometry, forced vital capacity (FVC), forced expiration volume in 1 second (FEV1), FEV1 / FVC ratio. Normal values of the FEV1 / FVC ratio between 0.7-0.8 and less than 0.65 are indicative of airway obstruction.
Number of hospitalizations | from baseline and at the end of the third months
  It shows the number of hospitalizations of the patient during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cross AJ, Thomas D, Liang J, Abramson MJ, George J, Zairina E. Educational interventions for health professionals managing chronic obstructive pulmonary disease in primary care. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012652. doi: 10.1002/14651858.CD012652.pub2. PMID 35514131
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549